CLINICAL TRIAL: NCT00949884
Title: A Randomized, Double-blind, Active-comparator, 8-week Forced-titration Study of the Efficacy and Safety of Olmesartan Medoxomil Versus Losartan Potassium in Hypertensive Subjects
Brief Title: Olmesartan Comparison to Losartan in Hypertensive Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Director, Medical Affairs, Daiichi Sankyo, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0866-A-U452
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Results first posted 2011-02-28 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olmesartan (Experimental): Olmesartan 20 mg once daily for four weeks followed by 40mg one daily for four weeks.
  Interventions: Drug: olmesartan medoxomil
- Placebo followed by Olmesartan (Placebo Comparator): Placebo capsule of olmesartan once daily for 2 weeks, followed by olmesartan 20 mg once daily for two weeks, followed by olmesartan 40 mg for 4 weeks
  Interventions: Drug: olmesartan medoxomil; Drug: Placebo
- Losartan (Active Comparator): Losartan 50 mg once daily for four weeks, followed by losartan 100 mg once daily for four weeks
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: olmesartan medoxomil — Oral tablets, once daily, at either 20mg or 40mg daily.
  Other Names: Benicar; Olmetec
  Arms: Olmesartan; Placebo followed by Olmesartan
Drug: Placebo — placebo oral tablets once daily for two weeks
  Arms: Placebo followed by Olmesartan
Drug: losartan potassium — losartan potassium oral tablet at either 50mg or 100 mg daily dose.
  Other Names: Cozaar
  Arms: Losartan

SUMMARY:
This study will evaluate the efficacy and safety of the FDA approved blood pressure medication olmesartan medoxomil compared to the FDA approved medication losartan potassium.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged > 18 years who are not institutionalized and have signed informed consent.
* Mean cuff seated diastolic blood pressure (BP) must be > 95 mmHg and < 115 mmHg and a mean cuff seated systolic BP must be < 180 mmHg when measured at two consecutive qualification study visits during the placebo run-in phase.
* The difference in mean cuff seated diastolic BP must be < 7 mmHg between two consecutive qualification study visits during the placebo run-in phase.

Exclusion Criteria:

* Subjects with type 2 diabetes mellitus with an HbA1c ≥ 9.5% at Screening.
* Subjects with serious disorders which may limit the ability to evaluate the efficacy or safety of olmesartan medoxomil and losartan potassium, including cardiovascular, renal (including the absence of one kidney), pulmonary, hepatic, gastrointestinal (including clinically significant malabsorption), endocrine/metabolic (with the exception of non-insulin, dependent type 2 diabetes mellitus with HbA1c < 9.5% at Screening), hematologic/oncologic (including an active malignancy other than basal cell carcinoma), neurologic and psychiatric diseases.
* Subjects with a history of myocardial infarction, angina, coronary angioplasty, bypass surgery or heart failure within the last 12 months.
* Subjects with any history of New York Heart Association Class III or IV congestive heart failure (CHF). A history of New York Heart Association Class I or II CHF may be exclusionary at the discretion of the Investigator.
* Subjects with a history of cerebrovascular accident or transient ischemic attack within the last 1 year.
* Subjects with clinically significant cardiac conduction defects, including second or third degree atrioventricular (AV) block, left bundle branch block, sick sinus syndrome, atrial fibrillation, atrial flutter, an accessory bypass tract, or any arrhythmia requiring medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Mesa, Arizona
  - Phoenix, Arizona
  - Harbor City, California
  - Tustin, California
  - Westlake Village, California
  - Pueblo, Colorado
  - Deerfield Beach, Florida
  - DeLand, Florida
  - South Bend, Indiana
  - Wichita, Kansas
  - Metairie, Louisiana
  - Albuquerque, New Mexico
  - Binghamton, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Greenville, South Carolina
  - Bristol, Tennessee
  - New Tazewell, Tennessee
  - Dallas, Texas
  - Norfolk, Virginia

REFERENCES:
- [Derived] Punzi HA, Lewin A, Li W, Chavanu KJ. Efficacy/safety of olmesartan medoxomil versus losartan potassium in naive versus previously treated subjects with hypertension. Adv Ther. 2012 Jun;29(6):524-37. doi: 10.1007/s12325-012-0029-5. Epub 2012 Jul 3. PMID 22763801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 119 out-patient centers throughout the U.S.: 1976 patients were screened, 1632 were enrolled, and 941 randomized.
Pre-assignment Details: Prior to group assignment was a 2-9 day screening period and a 3-4 week single-blind (participant was blinded) placebo run-in period. Participants were randomized in an 8:1:9 ratio to treatment arms as listed.
Period: Overall Study
Arm/Group | Olmesartan | Placebo Followed by Olmesartan | Losartan
Started | 420 | 52 | 469
Completed | 370 | 37 | 411
Not Completed | 50 | 15 | 58
Not completed — Adverse Event | 14 | 3 | 12
Not completed — Did not meet inclusion/exclusion | 2 | 1 | 3
Not completed — Lost to Follow-up | 7 | 5 | 5
Not completed — Physician Decision | 5 | 0 | 6
Not completed — Treatment non-compliance | 5 | 0 | 8
Not completed — Withdrawal by Subject | 13 | 4 | 16
Not completed — Lack of Efficacy | 4 | 2 | 7
Not completed — Study terminated by sponsor | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan | Placebo Followed by Olmesartan | Losartan | Total
Number analyzed (Participants) | 420 | 52 | 469 | 941
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 385 | 51 | 423 | 859
  >=65 years | 35 | 1 | 46 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (9.84) | 49.9 (8.67) | 52.1 (9.76) | 51.9 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 27 | 211 | 428
  Male | 230 | 25 | 258 | 513
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 7 | 61 | 120
  Not Hispanic or Latino | 368 | 45 | 408 | 821
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 2 | 6
  Asian | 25 | 2 | 26 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 118 | 16 | 133 | 267
  White | 273 | 33 | 304 | 610
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Hypertension stage [Number; unit: participants] — Hypertension stage was calculated using the baseline mean BP value. Stage I = systolic blood pressure of 140-159 mmHg and diastolic blood pressure 90-99 mmHg, Stage II = systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg
  participants
    Stage I | 120 | 23 | 134 | 277
    Stage II | 300 | 29 | 335 | 664
Height [Mean (Standard Deviation); unit: centimeter] | 169.92 (9.635) | 169.46 (9.652) | 170.47 (9.906) | 170.17 (9.767)
Weight [Mean (Standard Deviation); unit: kilogram] | 93.73 (19.627) | 96.14 (22.611) | 94.02 (21.647) | 94.01 (20.810)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter^2] | 32.41 (6.089) | 33.62 (8.103) | 32.28 (6.619) | 32.41 (6.480)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 158.3 (10.41) | 157.9 (10.05) | 158.3 (10.24) | 158.3 (10.29)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 101.1 (4.07) | 100.8 (3.79) | 101.3 (4.14) | 101.2 (4.09)
Pulse Rate [Mean (Standard Deviation); unit: beats per minute] | 78.8 (11.41) | 81.9 (9.88) | 78.5 (10.59) | 78.9 (10.94)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Trough, Cuff, Seated Diastolic Blood Pressure (SDBP)
Description: The change from baseline in trough SDBP at Week 8 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Day 0, Week 8
Population: The Efficacy Population included participants who received at least 1 dose of double-blind randomized study medication and had a baseline and at least 1 post-baseline blood pressure measurement. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Combined Olmesartan: Participants who were randomized to Olmesartan or to Placebo Followed by Olmesartan treatment arms, and received at least 1 high dose of olmesartan (40mg)
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 384 | 424 | 426
mmHg | -9.8 (0.50) | -9.7 (0.45) | -7.1 (0.45)
Statistical Analysis 1: Comparison: Combined Olmesartan vs Losartan; Null hypothesis was that there was no difference in change in seated diastolic blood pressure from baseline to end of treatment. Sample size of 900, this study had 90% power to detect a true difference in mean change from baseline in mean trough SDBP of 2.0 mmHg for Combined Olmesartan vs Losartan; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA model included treatment as a fixed effect and the baseline DBP as a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.8 to -1.3], Standard Error of Mean 0.63

2. Secondary Outcome: Change From Baseline to Week 4 in Trough, Cuff, Seated Systolic Blood Pressure (SSBP)
Description: The change from baseline in trough SSBP at Week 4 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Day 0, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 417 | 461 | 461
mmHg | -12.3 (0.67) | -12.0 (0.64) | -8.5 (0.64)
Statistical Analysis 1: Comparison: Combined Olmesartan vs Losartan; Test type: Superiority or Other; p < 0.0001, ANCOVA; The ANCOVA model included treatment as a fixed effect and baseline SSBP as a covariate; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-5.3 to -1.8], Standard Error of Mean 0.88

3. Secondary Outcome: Change From Baseline to Week 8 in Trough, Cuff, Seated Systolic Blood Pressure (SSBP)
Description: The change from baseline in trough SSBP at Week 8 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Day 0, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 384 | 424 | 426
mmHg | -13.6 (0.75) | -13.6 (0.71) | -9.7 (0.71)
Statistical Analysis 1: Comparison: Combined Olmesartan vs Losartan; Test type: Superiority or Other; p = 0.0001, ANCOVA; The ANCOVA model included treatment as a fixed effect and baseline SSBP as a covariate; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-5.8 to -1.9], Standard Error of Mean 0.99

4. Secondary Outcome: Change From Baseline to Week 4 in Trough, Cuff, Seated Diastolic Blood Pressure (SDBP)
Description: The change from baseline in trough SDBP at Week 4 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Day 0, Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 417 | 461 | 461
mmHg | -9.0 (0.44) | -8.8 (0.42) | -6.2 (0.42)
Statistical Analysis 1: Comparison: Combined Olmesartan vs Losartan; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included treatment as a fixed effect and baseline blood pressure value as a covariate; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-3.8 to -1.5], Standard Error of Mean 0.58

5. Post Hoc Outcome: Percentage of Participants Achieving Ambulatory Blood Pressure Goal of < 135/85 mmHg at Week 8
Description: Participants from pre-selected sites had 24-hour ambulatory blood pressure readings collected. Daytime readings were results collected between 8am and 4pm. Nighttime readings were results collected between 10pm and 6am.
Time Frame: Week 8
Population: Ambulatory Blood Pressure Monitoring (ABPM) Population: All participants in the Efficacy Population that had both valid (technically successful) baseline and Week 8 ambulatory blood pressure monitor data. A technically successful ABPM had at least 23 hours of ABPM data.
Measure: Number; unit: percentage of population
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 98 | 106 | 110
percentage of population
  Mean 24-hour | 59.2 | 58.5 | 40.9
  Mean Daytime | 32.7 | 32.1 | 21.8
  Mean Nighttime | 76.5 | 77.4 | 66.4

6. Other Pre Specified Outcome: Incremental Change From Week 4 to Week 8 in Trough, Cuff, Seated Diastolic Blood Pressure (SDBP)
Description: The change from Week 4 in trough SDBP at Week 8 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Week 4, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 384 | 424 | 426
mmHg | -0.8 (0.40) | -0.9 (0.38) | 0.0 (0.38)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Test type: Superiority or Other; p = 0.1121, ANCOVA; Treatment as a fixed effect and the seated cuff diastolic blood pressure value at week 4 (with last observation carried forward) as a covariate; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-2.0 to 0.2], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Test type: Superiority or Other; p = 0.0783, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-2.0 to 0.1], Standard Error of Mean 0.54

7. Other Pre Specified Outcome: Incremental Change From Week 4 to Week 8 in Trough, Cuff, Seated Systolic Blood Pressure (SSBP)
Description: The change from Week 4 in trough SSBP at Week 8 as measured by the Omron monitor. Morning doses of study medication were taken after the exam on study visit days, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Week 4, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 384 | 424 | 426
mmHg | -1.1 (0.66) | -1.4 (0.63) | 0.0 (0.63)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Test type: Superiority or Other; p = 0.2312, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.9 to 0.7], Standard Error of Mean 0.92
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Test type: Superiority or Other; p = 0.0979, ANCOVA; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.2 to 0.3], Standard Error of Mean 0.90

8. Other Pre Specified Outcome: Percentage of Participants Achieving Blood Pressure Goals at Week 4
Description: Percentage of participants who achieved the following goals:
  Systolic blood pressure: <140 mmHg, <135 mmHg, <130 mmHg, <120 mmHg Diastolic blood pressure: <90 mmHg, <85 mmHg, <80 mmHg Blood pressure: <140/90 mmHg, <135/80 mmHg, <130/80 mmHg
Time Frame: Week 4
Population: Efficacy population. Last observation carried forward. Denominator is the number of participants who have seated cuff BP measurement in each treatment group at any visit during the entire randomized treatment phase. Participants randomized to placebo-olmesartan, the measurement is after at least one dose of olmesartan.
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 417 | 461 | 461
percentage of participants analyzed
  Systolic BP <140 mmHg | 37.9 | 36.7 | 25.6
  Systolic BP <135 mmHg | 28.1 | 27.1 | 14.1
  Systolic BP <130 mmHg | 16.8 | 16.5 | 7.2
  Systolic BP <120 mmHg | 3.1 | 3.5 | 2.0
  Diastolic BP <90 mmHg | 39.6 | 38.8 | 24.5
  Diastolic BP <85 mmHg | 24.2 | 23.9 | 13.0
  Diastolic BP <80 mmHg | 10.6 | 10.4 | 4.6
  Blood pressure <140/90 mmHg | 27.3 | 26.5 | 14.3
  Blood pressure <135/80 mmHg | 7.4 | 7.6 | 2.2
  Blood pressure <130/80 mmHg | 5.5 | 5.9 | 1.5
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <140 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <140 mmHg; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <135 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <135 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <130 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 6: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <130 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <120 mmHg; Test type: Superiority or Other; p = 0.2755, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <120 mmHg; Test type: Superiority or Other; p = 0.1646, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 9: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 10: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 11: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <85 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 12: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <85 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 13: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <80 mmHg; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 14: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <80 mmHg; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 15: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <140/90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 16: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <140/90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 17: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <135/80 mmHg; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 18: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <135/80 mmHg; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 19: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <130/80 mmHg; Test type: Superiority or Other; p = 0.0023, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 20: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <130/80 mmHg; Test type: Superiority or Other; p = 0.0012, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates

9. Other Pre Specified Outcome: Percentage of Participants Achieving Blood Pressure Goals at Week 8
Description: Percentage of participants who achieved the following goals:
  Systolic blood pressure: <140 mmHg, <135 mmHg, <130 mmHg, <120 mmHg Diastolic blood pressure: <90 mmHg, <85 mmHg, <80 mmHg Blood pressure: <140/90 mmHg, <135/80 mmHg, <130/80 mmHg, <120/80 mmHg
Time Frame: Week 8
Population: as for outcome 8
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 384 | 424 | 426
percentage of participants analyzed
  Systolic BP <140 mmHg | 41.1 | 41.0 | 28.9
  Systolic BP <135 mmHg | 29.9 | 30.0 | 20.4
  Systolic BP <130 mmHg | 18.2 | 18.4 | 13.1
  Systolic BP <120 mmHg | 6.8 | 6.6 | 3.8
  Diastolic BP <90 mmHg | 43.2 | 42.5 | 30.5
  Diastolic BP <85 mmHg | 22.9 | 22.9 | 15.5
  Diastolic BP <80 mmHg | 12.2 | 11.8 | 6.6
  Blood pressure <140/90 mmHg | 32.6 | 31.6 | 19.5
  Blood pressure <135/80 mmHg | 10.2 | 9.9 | 4.9
  Blood pressure <130/80 mmHg | 7.6 | 7.5 | 4.5
  Blood pressure <120/80 mmHg | 4.9 | 4.7 | 2.3
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <140 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <140 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <135 mmHg; Test type: Superiority or Other; p = 0.0009, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <135 mmHg; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <130 mmHg; Test type: Superiority or Other; p = 0.0347, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 6: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <130 mmHg; Test type: Superiority or Other; p = 0.0280, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <120 mmHg; Test type: Superiority or Other; p = 0.0519, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving systolic blood pressure goal of <120 mmHg; Test type: Superiority or Other; p = 0.0605, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 9: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <90 mmHg; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 10: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <90 mmHg; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 11: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <85 mmHg; Test type: Superiority or Other; p = 0.0070, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 12: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <85 mmHg; Test type: Superiority or Other; p = 0.0066, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 13: Comparison: Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <80 mmHg; Test type: Superiority or Other; p = 0.0061, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 14: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving diastolic blood pressure goal of <80 mmHg; Test type: Superiority or Other; p = 0.0096, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 15: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <140/90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 16: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <140/90 mmHg; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 17: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <135/80 mmHg; Test type: Superiority or Other; p = 0.0047, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 18: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <135/80 mmHg; Test type: Superiority or Other; p = 0.0063, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 19: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <130/80 mmHg; Test type: Superiority or Other; p = 0.0589, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 20: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <130/80 mmHg; Test type: Superiority or Other; p = 0.0594, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 21: Comparison: Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <120/80 mmHg; Test type: Superiority or Other; p = 0.0476, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates
Statistical Analysis 22: Comparison: Combined Olmesartan vs Losartan; Percentage of participants achieving blood pressure goal of <120/80 mmHg; Test type: Superiority or Other; p = 0.0657, Regression, Logistic; The p-value is from the logistic regression with treatment as the main effect and baseline SSBP or SDBP as covariates

10. Other Pre Specified Outcome: Change From Baseline in Mean 24-Hour Ambulatory Blood Pressure at Week 4
Description: In week 4, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours.
Time Frame: Baseline, Week 4
Population: The ABPM population was defined as all participants in the efficacy population that had valid (technically successful required at least 23 hours of ABPM data) baseline and Week 4 ABPM data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 108 | 118 | 118
mmHg
  Systolic blood pressure | -7.3 (1.08) | -7.3 (1.03) | -5.9 (1.03)
  Diastolic blood pressure | -4.9 (0.70) | -4.8 (0.67) | -3.7 (0.67)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Change from baseline at week 4 in systolic blood pressure; Test type: Superiority or Other; p = 0.3250, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure as a covariate; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.4 to 1.5]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Change from baseline at week 4 in systolic blood pressure; Test type: Superiority or Other; p = 0.3491, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure as a covariate; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-4.4 to 1.5]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Change from baseline at week 4 in diastolic blood pressure; Test type: Superiority or Other; p = 0.2085, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.2 to 0.7]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Change from baseline at week 4 in diastolic blood pressure; Test type: Superiority or Other; p = 0.2542, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.0 to 0.8]

11. Other Pre Specified Outcome: Change From Baseline in Mean 24-Hour Ambulatory Blood Pressure at Week 8
Description: In week 8, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours.
Time Frame: Baseline, Week 8
Population: The ABPM population was defined as all participants in the efficacy population that had valid (technically successful required at least 23 hours of ABPM data) baseline and Week 8 ABPM data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 98 | 106 | 110
mmHg
  Systolic blood pressure | -9.1 (1.16) | -9.2 (1.11) | -5.6 (1.09)
  Diastolic blood pressure | -6.1 (0.78) | -6.1 (0.75) | -3.6 (0.73)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Change from baseline at week 8 in systolic blood pressure; Test type: Superiority or Other; p = 0.0209, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-6.6 to -0.5]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Change from baseline at week 8 in systolic blood pressure; Test type: Superiority or Other; p = 0.0186, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-6.6 to -0.6]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Change from baseline at week 8 in diastolic blood pressure; Test type: Superiority or Other; p = 0.0175, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.5 to -0.4]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Change from baseline at week 8 in diastolic blood pressure; Test type: Superiority or Other; p = 0.0177, ANCOVA; Treatment is a fixed effect and baseline mean 24-hour ABPM blood pressure is a covariate; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.4 to -0.4]

12. Other Pre Specified Outcome: Change From Baseline in Mean Daytime (8am to 4pm) and Mean Nighttime (10pm to 6am) Ambulatory Blood Pressure at Week 4
Description: In week 4, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours. Daytime (8am to 4pm) and nighttime (10pm to 6am) systolic and diastolic blood pressure readings are summarized.
Time Frame: Baseline, Week 4
Population: The ambulatory blood pressure monitor (ABPM) population was defined as participants in the efficacy population that had valid baseline and Week 4 ABPM data. Valid (technically successful) ABPM had at least 23 hours of ABPM data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 108 | 118 | 118
mmHg
  Daytime systolic blood pressure | -7.6 (1.27) | -7.5 (1.22) | -5.8 (1.22)
  Daytime diastolic blood pressure | -5.4 (0.84) | -5.2 (0.81) | -3.5 (0.81)
  Nighttime systolic blood pressure | -6.7 (1.15) | -6.8 (1.10) | -5.5 (1.10)
  Nighttime diastolic blood pressure | -4.4 (0.77) | -4.3 (0.74) | -3.4 (0.74)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Daytime systolic blood pressure; Test type: Superiority or Other; p = 0.3104, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.2 to 1.7]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Daytime systolic blood pressure; Test type: Superiority or Other; p = 0.3653, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-4.9 to 1.8]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Daytime diastolic blood pressure; Test type: Superiority or Other; p = 0.1197, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.1 to 0.5]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Daytime diastolic blood pressure; Test type: Superiority or Other; p = 0.1654, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.9 to 0.7]
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; Nighttime systolic blood pressure; Test type: Superiority or Other; p = 0.4362, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-4.4 to 1.9]
Statistical Analysis 6: Comparison: Combined Olmesartan vs Losartan; Nighttime systolic blood pressure; Test type: Superiority or Other; p = 0.4039, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-4.5 to 1.8]
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; Nighttime diastolic blood pressure; Test type: Superiority or Other; p = 0.3929, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.1 to 1.2]
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; Nighttime diastolic blood pressure; Test type: Superiority or Other; p = 0.4259, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.0 to 1.3]

13. Other Pre Specified Outcome: Change From Baseline in Mean Daytime (8am to 4pm) and Mean Nighttime (10pm to 6am) Ambulatory Blood Pressure at Week 8
Description: In week 8, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours. Daytime (8am to 4pm) and nighttime (10pm to 6am) systolic and diastolic blood pressure readings are summarized.
Time Frame: Baseline, Week 8
Population: The ambulatory blood pressure monitor (ABPM) population was defined as participants in the efficacy population that had valid baseline and Week 8 ABPM data. Valid (technically successful) ABPM had at least 23 hours of ABPM data.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 98 | 106 | 110
mmHg
  Daytime systolic blood pressure | -8.7 (1.24) | -8.7 (1.20) | -5.2 (1.17)
  Daytime diastolic blood pressure | -6.2 (0.86) | -6.1 (0.83) | -3.7 (0.82)
  Nighttime systolic blood pressure | -9.3 (1.32) | -9.3 (1.27) | -6.3 (1.25)
  Nighttime diastolic blood pressure | -6.2 (0.91) | -6.1 (0.87) | -4.1 (0.86)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; Daytime systolic blood pressure; Test type: Superiority or Other; p = 0.0396, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.8 to -0.2]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; Daytime systolic blood pressure; Test type: Superiority or Other; p = 0.0345, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-6.8 to -0.3]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; Daytime diastolic blood pressure; Test type: Superiority or Other; p = 0.0324, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-4.8 to -0.2]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; Daytime diastolic blood pressure; Test type: Superiority or Other; p = 0.0363, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.7 to -0.2]
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; Nighttime systolic blood pressure; Test type: Superiority or Other; p = 0.0988, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.5 to 0.6]
Statistical Analysis 6: Comparison: Combined Olmesartan; Nighttime systolic blood pressure; Test type: Superiority or Other; p = 0.0926, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-6.4 to 0.5]
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; Nighttime diastolic blood pressure; Test type: Superiority or Other; p = 0.0900, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-4.5 to 0.3]
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; Nighttime diastolic blood pressure; Test type: Superiority or Other; p = 0.0942, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.4 to 0.3]

14. Other Pre Specified Outcome: Change From Baseline in Mean Ambulatory Blood Pressure During the Final 2, 4, and 6 Hours of the Dosing Interval at Week 4
Description: In week 4, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours. Systolic and diastolic blood pressure readings taken in the final 2, 4, and 6 hours of the 24-hour ABPM cycle are summarized.
Time Frame: Baseline, Week 4
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 108 | 118 | 118
mmHg
  2 hour systolic blood pressure | -8.7 (1.31) | -8.4 (1.26) | -6.8 (1.26)
  2 hour diastolic blood pressure | -5.8 (0.94) | -5.6 (0.90) | -3.8 (0.90)
  4 hour systolic blood pressure | -8.4 (1.23) | -8.3 (1.18) | -6.5 (1.18)
  4 hour diastolic blood pressure | -5.8 (0.85) | -5.6 (0.82) | -4.1 (0.82)
  6 hour systolic blood pressure | -8.0 (1.18) | -8.0 (1.13) | -6.2 (1.13)
  6 hour diastolic blood pressure | -5.5 (0.83) | -5.4 (0.79) | -3.9 (0.79)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; 2 hour systolic blood pressure; Test type: Superiority or Other; p = 0.3229, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.4 to 1.8]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; 2 hour systolic blood pressure; Test type: Superiority or Other; p = 0.3863, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-5.1 to 2.0]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; 2 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1277, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.5 to 0.6]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; 2 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1799, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-4.3 to 0.8]
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; 4 hour systolic blood pressure; Test type: Superiority or Other; p = 0.2708, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.1 to 1.4]
Statistical Analysis 6: Comparison: Combined Olmesartan vs Losartan; 4 hour systolic blood pressure; Test type: Superiority or Other; p = 0.3133, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-5.0 to 1.6]
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; 4 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1621, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.9 to 0.7]
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; 4 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.2314, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.7 to 0.9]
Statistical Analysis 9: Comparison: Olmesartan vs Losartan; 6 hour systolic blood pressure; Test type: Superiority or Other; p = 0.2461, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-5.0 to 1.3]
Statistical Analysis 10: Comparison: Combined Olmesartan vs Losartan; 6 hour systolic blood pressure; Test type: Superiority or Other; p = 0.2558, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-5.0 to 1.3]
Statistical Analysis 11: Comparison: Olmesartan vs Losartan; 6 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1700, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.8 to 0.7]
Statistical Analysis 12: Comparison: Combined Olmesartan vs Losartan; 6 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.2011, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-3.7 to 0.8]

15. Other Pre Specified Outcome: Change From Baseline in Mean Ambulatory Blood Pressure During the Final 2, 4, and 6 Hours of the Dosing Interval at Week 8
Description: In week 8, participants arrived at the site in the morning without having taken that day's dose of medication. Once the ambulatory blood pressure monitor (ABPM) had been applied, medication was taken and the participant wore the ABPM for a period of 24-hours. Systolic and diastolic blood pressure readings taken in the final 2, 4, and 6 hours of the 24-hour ABPM cycle are summarized.
Time Frame: Baseline, Week 8
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Combined Olmesartan | Losartan
Number analyzed (Participants) | 98 | 106 | 110
mmHg
  2 hour systolic blood pressure | -10.0 (1.56) | -9.5 (1.50) | -7.2 (1.48)
  2 hour diastolic blood pressure | -6.3 (1.10) | -6.0 (1.06) | -4.0 (1.04)
  4 hour systolic blood pressure | -10.5 (1.40) | -10.1 (1.35) | -6.9 (1.32)
  4 hour diastolic blood pressure | -7.1 (0.96) | -6.7 (0.93) | -4.1 (0.91)
  6 hour systolic blood pressure | -10.0 (1.33) | -9.7 (1.28) | -6.5 (1.25)
  6 hour diastolic blood pressure | -6.8 (0.92) | -6.5 (0.89) | -4.0 (0.87)
Statistical Analysis 1: Comparison: Olmesartan vs Losartan; 2 hour systolic blood pressure; Test type: Superiority or Other; p = 0.1895, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-7.0 to 1.4]
Statistical Analysis 2: Comparison: Combined Olmesartan vs Losartan; 2 hour systolic blood pressure; Test type: Superiority or Other; p = 0.2701, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-6.5 to 1.8]
Statistical Analysis 3: Comparison: Olmesartan vs Losartan; 2 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1328, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-5.2 to 0.7]
Statistical Analysis 4: Comparison: Combined Olmesartan vs Losartan; 2 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.1778, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-4.9 to 0.9]
Statistical Analysis 5: Comparison: Olmesartan vs Losartan; 4 hour systolic blood pressure; Test type: Superiority or Other; p = 0.0620, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.6, 95% CI 2-sided [-7.3 to 0.2]
Statistical Analysis 6: Comparison: Combined Olmesartan vs Losartan; 4 hour systolic blood pressure; Test type: Superiority or Other; p = 0.1011, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-6.9 to 0.6]
Statistical Analysis 7: Comparison: Olmesartan vs Losartan; 4 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.0249, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-5.6 to -0.4]
Statistical Analysis 8: Comparison: Combined Olmesartan vs Losartan; 4 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.0497, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-5.2 to 0.0]
Statistical Analysis 9: Comparison: Olmesartan vs Losartan; 6 hour systolic blood pressure; Test type: Superiority or Other; p = 0.0552, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-7.1 to 0.1]
Statistical Analysis 10: Comparison: Combined Olmesartan vs Losartan; 6 hour systolic blood pressure; Test type: Superiority or Other; p = 0.0767, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-6.8 to 0.3]
Statistical Analysis 11: Comparison: Olmesartan vs Losartan; 6 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.0279, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-5.3 to -0.3]
Statistical Analysis 12: Comparison: Combined Olmesartan vs Losartan; 6 hour diastolic blood pressure; Test type: Superiority or Other; p = 0.0434, ANCOVA; Treatment was a fixed effect and baseline mean daytime and nighttime ABPM blood pressure was a covariate; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.0 to -0.1]

16. Other Pre Specified Outcome: Change From Baseline to Week 2 in Trough, Cuff, Seated Blood Pressure
Description: The change from baseline in trough systolic and diastolic blood pressure at Week 2 as measured by the Omron monitor. Morning doses of study medication were taken after the exam, therefore exam measurements were taken when medication levels were at its lowest ('the trough'). Following a 5-minute rest period, three separate blood pressure measurements were taken with a full 2-minute (not exceeding 5 minutes) interval between measurements, with the cuff fully deflated between measurements. The mean of the 3 seated blood pressure measurements constitute the blood pressure value for the visit.
Time Frame: Baseline, Week 2
Population: The efficacy population was defined as participants who received at least 1 dose of double-blind randomized study medication and had a baseline and at least 1 post-baseline blood pressure measurement. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Olmesartan | Placebo Followed by Olmesartan | Losartan
Number analyzed (Participants) | 417 | 50 | 0
mmHg
  Diastolic blood pressure | -8.3 (0.42) | -4.0 (1.22) |
  Systolic blood pressure | -11.9 (0.65) | -3.3 (1.87) |
Statistical Analysis 1: Comparison: Olmesartan vs Placebo Followed by Olmesartan; Diastolic blood pressure; Test type: Superiority or Other; p = 0.0009, ANCOVA; Treatment is a fixed effect and baseline blood pressure is a covariate; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-6.8 to -1.8]
Statistical Analysis 2: Comparison: Olmesartan vs Placebo Followed by Olmesartan; Systolic blood pressure; Test type: Superiority or Other; p < 0.0001, ANCOVA; Treatment is a fixed effect and baseline blood pressure is a covariate; Mean Difference (Final Values) = -8.6, 95% CI 2-sided [-12.5 to -4.7]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 8, or until the adverse event resolved or the condition stabilized.
Description: Safety population includes all participants who received at least 1 dose of double-blind randomized study medication
Arm/Group | Olmesartan | Placebo Followed by Olmesartan | Losartan
Serious Adverse Events (participants affected / at risk) | 0/420 | 0/52 | 4/469
Other Adverse Events (participants affected / at risk) | 133/420 | 21/52 | 148/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan (N=420) | Placebo Followed by Olmesartan (N=52) | Losartan (N=469)
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cerebrovasular accident (Nervous system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan (N=420) | Placebo Followed by Olmesartan (N=52) | Losartan (N=469)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 4
Type II hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 3
Diplopia (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 2 | 9
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 4
Feeling cold (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 3
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 6 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cutaneous larva migrans (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 1
Influenza (Infections and infestations) | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 8 | 0 | 13
Oral fungal infection (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 3
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 10
Urinary tract infection (Infections and infestations) | 4 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatinine abnormal (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1
Blood sodium increased (Investigations) | 1 | 1 | 2
Blood triglycerides increased (Investigations) | 2 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 1
Liver function test abnormal (Investigations) | 2 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 1
Lymphocyte morphology abnormal (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 8 | 1 | 6
Headache (Nervous system disorders) | 18 | 5 | 24
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 3
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Dysthymic disorder (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 4
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 1 | 4
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reflects the following restrictive language in the Clinical Study Agreements: "If identified by DSI, any of DSI's confidential information as defined herein shall be deleted…Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by the Study Site."